CLINICAL TRIAL: NCT02992236
Title: Effects of the NO-synthase Inhibitor VAS203 on Renal Function in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: veriNOS operations GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: VAS203/I/3/05
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Renal Function Impairment in Healthy Volunteers
MeSH Terms: interventions — 4-amino-tetrahydrobiopterin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Infusion (6 hours) of Saline
  Interventions: Drug: Saline
- VAS203 (Active Comparator): Infusion (6 hours) of VAS203 (10 mg/kg)
  Interventions: Drug: VAS203

INTERVENTIONS:
Drug: VAS203 — Infusion of NO-Synthase inhibitor VAS203
  Other Names: Ronopterin
  Arms: VAS203
Drug: Saline — Infusion of saline
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Analysis of the effect of the NO-Synthase inhibitor VAS203 (6 hours infusion of 10 mg/kg) on renal function and perfusion in 16 healthy subjects.

DETAILED DESCRIPTION:
Analysis of the effect of i.v. VAS203 on renal function and perfusion in healthy subjects.

Primary objective:

Possible adverse effect of VAS203 on the Renal Plasma Flow (RPF) and the Glomerular Filtration Rate (GFR) during and after 6 hours of constant-rate iv. infusion of 10 mg/kg VAS203.

Secondary objective:

To analyse the effects of VAS203 on

* filtration fraction
* hemodynamics (afferent and efferent resistance, intraglomerular pressure)
* markers of kidney injury and renal function
* systolic, mean and diastolic brachial blood pressure
* Plasma Pharmacokinetic of VAS203 and its first metabolite.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent in writing available.
2. Willing and able to comply with all requirements of the study.
3. Male, 18 and 45 years (inclusive).
4. Subject has a body weight between 60 kg and 100 kg, extremes included.
5. BMI 18 to 27 kg/m2.
6. Non-smoker
7. Serum creatinine within reference range (≤1.2 mg/dL) and Cockroft-Gault Clearance > 90 ml/min
8. Good general health as judged by the Investigator, as determined by medical history, physical examination, vital signs (systolic and diastolic blood pressure and pulse rate) and clinical laboratory parameters (clinical chemistry, hematology, and urinalysis)

Exclusion Criteria:

1. Clinically significant abnormalities in physical examination, vital signs or clinical laboratory parameters (according to the Investigator's judgment).
2. Serum glutamate oxaloacetate transaminase or glutamate-pyruvate transaminase > 2-times above the upper limit of normal range.
3. Subject with Cockcroft-Gault clearance < 90 ml/min.
4. Clinically significant history of cardiovascular disease or any known present cardiovascular disease.
5. History of clinically significant neurological, gastrointestinal, renal, hepatic, psychological, pulmonary, metabolic, endocrine, hematological, or other major disorders.
6. Office blood pressure at screening higher than 160/100 mmHg, or lower than 95/55 mmHg.
7. Office heart rate at screening after at least 5 minutes outside the range of 50- 99 beats per minute (inclusive).
8. Concomitant use of OTC medication within 1 week prior to dosing, except use of paracetamol (up to 2 g/day).
9. Participation in any other clinical study within 30 days prior to inclusion in this -

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Prof. Dr., Principal Investigator — Universitätsklinik Erlangen
Locations (1):
- Universitätsklinik Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cross-over design, all subjects received VAS203 and placebo
Groups:
- Placebo, Then VAS203: Participants first received Placebo (6 hours Infusion of Saline). After a washout period of 4 weeks, they then received VAS203 (6 hours Infusion of 10 mg/kg VAS203).
- VAS203, Then Placebo: Participants first received VAS203 (6 hours Infusion of 10 mg/kg VAS203). After a washout period of 4 weeks, they then received Placebo (6 hours Infusion of Saline).
Period: Overall Study
Arm/Group | Placebo, Then VAS203 | VAS203, Then Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then VAS203 | VAS203, Then Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (7.9) | 31.2 (7.9) | 31.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Germany | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Renal Plasma Flow
Description: Renal plasma flow measurement by para-Amino-Hippuric-Acid Clearance Method
Time Frame: 0, 2h, 4h, 6h and 8 h after start of infusion
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo | VAS203
Number analyzed (Participants) | 16 | 16
mL/min | 541 (85) | 663 (125)
Statistical Analysis 1: Comparison: Placebo vs VAS203; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Primary Outcome: Glomerular Filtration Rate
Description: by para-Amino-Hippuric Acid Clearance Method
Time Frame: 0, 2h, 4h, 6h and 8 h after start of infusion
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- VAS203: Six hours infusion of 10 mg/kg VAS203.
- Placebo: Six hours Infusion of Saline
Arm/Group | VAS203 | Placebo
Number analyzed (Participants) | 16 | 16
mL/min | 135 (15) | 153.5 (15)

3. Secondary Outcome: Serum Creatinine Concentration
Time Frame: 0, 2h, 4h, 6h, 8h, 10h, 24h and 48h after start of infusion
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | VAS203
Number analyzed (Participants) | 16 | 16
mg/dL | 0.91 (0.1) | 0.94 (0.1)

ADVERSE EVENTS:
Arm/Group | Placebo | VAS203
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | VAS203 (N=16)
Headache (Nervous system disorders) | 1 (1) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No